CLINICAL TRIAL: NCT05450185
Title: The Effect of Filter Lifespan in Continuous Renal Replacement Therapy on the Rate of New Infections in Critically Ill Patients: a Prospective, Multicenter, Observational Trial
Brief Title: Filter Lifespan in Continuous Renal Replacement Therapy
Acronym: CRRTInfO
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-AnIt-21
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Critically Ill; Continuous Renal Replacement Therapy; Infections
MeSH Terms: conditions — Critical Illness; Infections | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma, urine, dialysate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Critically ill patients with continuous renal replacement therapy — Due to the observational design of the study, no study-specific interventions are performed. The treatment of the patients is completely guided by the responsible ICU physicians.

SUMMARY:
The only supportive therapy for patients with AKI is renal replacement therapy (RRT). In the ICU setting, continuous RRT (CRRT) is mostly favored. In a post-hoc analysis of the RICH trial (regional citrate versus systemic heparin anticoagulation for CRRT in critically ill patient with AKI), it was shown that the filter life span is associated with an increased rate of new infection and that the type of anticoagulants did not directly affect infection rate. The mechanisms of this infection rate is unknown.

DETAILED DESCRIPTION:
Approximately every second patient in the ICU suffers from acute kidney injury (AKI) which complicates the clinical course of these patients. Continuous renal replacement therapy (CRRT) has become the most widely used form of renal support in critically ill patients as it allows continuous, controlled removal of fluids and is hemodynamically better tolerated compared to intermittent dialysis. The requirement for intravascular access and artificial circuits may increase the risk of infection. However, there are no studies analyzing the incidence and characteristics of infections in critically ill patients with CRRT or the implications for outcome. Therefore, this observational trial investigates the factors that influences new onset infection in critically ill patients with CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Critically ill patients with dialysis-dependent AKI
* Continuous renal replacement therapy (CRRT)
* Written informed consent

Exclusion Criteria:

* Chronic kidney disease with estimated glomerular filtration rate (eGFR)<30ml/min/1.73m2
* Chronic dialysis dependency
* Kidney transplant
* (Glomerulo-)nephritis, interstitial nephritis, vasculitis
* Patients on immunosuppression
* Patients with chronic inflammatory diseases (e.g. arthritis, HIV, chronic hepatitis)
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of new infections since start of dialysis | From start of dialysis until day 28

SECONDARY OUTCOMES:
Number of new blood stream infections | From start of dialysis until day 28
Number of new pneumonia | From start of dialysis until day 28
Number of new urinary tract infection | From start of dialysis until day 28
Number of new catheter blood stream infection | From start of dialysis until day 28
Number of new other infections | From start of dialysis until day 28
Filter live span | From start of dialysis until day 28 or end of CRRT, whatever occurs first
Number of bacterial contamination of t he CRRT circuit proven by culture | From start of dialysis until day 28 or end of CRRT, whatever occurs first
Down-time of CRRT in hours | From start of dialysis until day 28 or end of CRRT, whatever occurs first
Days on renal replacement therapy | From start of dialysis until day 28
Duration of mechanical ventilation in hours | From start of dialysis until day 28
Number of bleeding complications | From start of dialysis until day 28
  defined as bleeding with the need for at least 1 packed red cells (RBC)
Recovery of kidney function | At day 28 after start of dialysis
  Recovery of kidney function (defined as complete recovery: serum-creatinine ≤0.5 mg/dl higher than baseline; partial recovery: serum creatinine >0.5 mg/dl higher than baseline but no dialysis-dependence; non-recovery: patients who remained dialysis-dependent)
Recovery of kidney function | At day 60 after start of dialysis
  Recovery of kidney function (defined as complete recovery: serum-creatinine ≤0.5 mg/dl higher than baseline; partial recovery: serum creatinine >0.5 mg/dl higher than baseline but no dialysis-dependence; non-recovery: patients who remained dialysis-dependent)
Recovery of kidney function | At day 90 after start of dialysis
  Recovery of kidney function (defined as complete recovery: serum-creatinine ≤0.5 mg/dl higher than baseline; partial recovery: serum creatinine >0.5 mg/dl higher than baseline but no dialysis-dependence; non-recovery: patients who remained dialysis-dependent)
Number of patients with need for kidney replacement therapy | At day 28 after start of dialysis
Number of patients with need for kidney replacement therapy | At day 60 after start of dialysis
Number of patients with need for kidney replacement therapy | At day 90 after start of dialysis
Mortality | At day 28 after start of dialysis
Mortality | At day 60 after start of dialysis
Mortality | At day 90 after start of dialysis
Major adverse kidney events (MAKE) | At day 28 after start of dialysis
  Composite endpoint consisting of death, renal replacement therapy, and persistent renal dysfunction
Major adverse kidney events (MAKE) | At day 60 after start of dialysis
  Composite endpoint consisting of death, renal replacement therapy, and persistent renal dysfunction
Major adverse kidney events (MAKE) | At day 90 after start of dialysis
  Composite endpoint consisting of death, renal replacement therapy, and persistent renal dysfunction

OTHER OUTCOMES:
Transmigration of neutrophils | At initiation of dialysis
Transmigration of neutrophils | 24 hours after initiation of dialysis
Transmigration of neutrophils | 48 hours after initiation of dialysis
Transmigration of neutrophils | 72 hours after initiation of dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Principal Investigator — University Hospital Münster
Locations (5):
- Univ.-Klinik Innsbruck, Innsbruck, Austria
- Universidade de São Paulo, São Paulo, Brazil
- Germany (3):
  - Universitätsklinikum Erlangen-Nürnberg, Abteilung für Nephrologie und Hypertensiologie, Erlangen
  - Kliniken Maria Hilf, Klinik für Anästhesiologie und Operative Intensivmedizin, Mönchengladbach
  - University Hospital Muenster, Münster